CLINICAL TRIAL: NCT01485146
Title: A Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ETC-1002 at Doses Above 120 mg/Day in Healthy Subjects
Brief Title: A Multiple Ascending Dose Study of ETC-1002 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ETC-1002-004
Record Dates: First submitted 2011-10-25; First posted 2011-12-05 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Safety Evaluation of Escalating Doses
MeSH Terms: interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): 8 Healthy Subjects in Phase I Unit
  Interventions: Drug: ETC-1002
- Cohort 2 (Experimental): 8 Healthy Subjects in Phase I Unit
  Interventions: Drug: ETC-1002
- Cohort 3 (Experimental): 8 Healthy Subjects in Phase I Unit
  Interventions: Drug: ETC-1002

INTERVENTIONS:
Drug: ETC-1002 — escalating doses

SUMMARY:
This Phase 1, double-blind (sponsor open), placebo controlled study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of ETC-1002 in healthy subjects.

ELIGIBILITY:
Major Inclusion Criteria:

* Healthy male and female subjects of non-child bearing potential as determined by medical history, physical exam and vial sign measurements
* Body Mass Index of 18-32 kg/m2 inclusive with body weight >50 kg

Major Exclusion Criteria:

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.2 x Upper Limit of Normal(ULN), serum creatinine >ULN, Hemoglobin <12.0 g/dL
* Clinically significant disease that requires a physician's care and/or would interfere with study evaluations
* History of drug or alcohol abuse, consumption of alcohol within 48 hours prior to randomization, or a positive test for alcohol or drugs with a high potential for abuse prior to randomization
* Use of any prescription or nonprescription drugs, vitamins, or dietary supplements within 14 days prior to randomization
* Other exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2012-01-25 (Actual); Study Completion 2012-01-25 (Actual)

PRIMARY OUTCOMES:
Measuring subject safety by collecting and evaluating vital signs, adverse events, and laboratory measures. | 14 days

SECONDARY OUTCOMES:
Measuring the level of ETC-1002 and its metabolite ESP15228 in the blood. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Lalwani, PhD, Study Director — Esperion Therapeutics, Inc.
Locations (1):
- Jasper Clinic, Inc., Kalamazoo, Michigan, United States